CLINICAL TRIAL: NCT05676515
Title: Evaluation of Different Culture Media for in Vitro Fertilization: a Randomized Clinical Trial
Brief Title: Evaluation of Different Culture Media for in Vitro Fertilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Guedes da Luz Médicos Associados Sociedade Simples LTDA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 60500922.2.0000.5327
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Infertility, Female
Keywords: culture media; fertilization
MeSH Terms: conditions — Infertility, Female | interventions — Culture Media

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- culture media of fabricant A (Active Comparator): use of culture media of fabricant A
  Interventions: Other: culture media
- culture media of fabricant B (Active Comparator): use of culture media of fabricant B
  Interventions: Other: culture media
- culture media of fabricant C (Active Comparator): use of culture media of fabricant C
  Interventions: Other: culture media

INTERVENTIONS:
Other: culture media — spliting of biological material and use of three culture media

SUMMARY:
Under in vivo conditions, human gametes and embryos are exposed to fluids in the fallopian tubes, where fertilization occurs, and in the uterus, the site of embryonic implantation. The composition of these microenvironments is extremely complex and diverse. On the other hand, infertile couples who need in vitro fertilization treatments have their gametes and embryos cultured for a few days in commercial culture media. The composition of the media used in assisted reproduction laboratories varies according to the manufacturer and culture strategy. It is already known that the exposure of embryos to different concentrations of nutrients can affect the effectiveness of in vitro fertilization treatments, such as the fertilization rate, embryonic development speed, implantation rate, gestation, abortion, newborn weight, among other factors. Although these aspects are much discussed in the literature, there is still no consensus regarding the choice of a specific culture medium. Thus, the present study aims to evaluate the influence of three commercial culture media on the fertilization rate and embryonic quality through a prospective randomized clinical trial using sibling oocytes from patients undergoing in vitro fertilization cycles.

DETAILED DESCRIPTION:
For this prospective randomized clinical trial, patients undergoing IVF cycles with at least three oocytes obtained from ovarian aspiration procedure will be enrolled. Considering a 30% difference between the groups in the number of good quality embryos (A + B) with power of 80% and p alpha 5%, the n calculated was 95 oocytes for each group, totaling 285 oocytes retrieved and 48 patients, as the mean number of oocytes per patient is 6.

The two main parameters that will be evaluated are:

Fertilization rate: An oocyte with 2 pronuclei and 2 polar bodies formed (2PN/2CPs) is considered fertilized. The evaluation of oocyte fertilization rates in three tested media will be measured by the percentage of 2PN/2CPs zygotes observed in the check between 16-18 hours after fertilization by IVF or ICSI.

Embryo quality: Embryos will be classified as A, B, C or D according to the scheme below, with A and B embryos being considered good quality embryos. The evaluation of embryonic quality will be carried out on the third day (64-67 hours after fertilization) taking into account the parameters of cell number, symmetry and fragmentation.

Embryo quality was defined as the primary outcome of this study because it is a parameter directly related to the prognosis of in vitro fertilization treatment, and it has a predefined value in the Vienna consensus being commonly described in scientific articles.

Fertilization rates and good quality embryos will be expressed as percentages (mean and standard deviation). The chi-square test will be used to compare fertilization and embryonic quality between the culture media and the difference will be considered significant if p < 0.05. For tabulation and statistical analysis, the JASP software version 0.16.2 will be used.

ELIGIBILITY:
Inclusion Criteria:

* IVF/ICSI cycles;
* At least three oocytes retrieved;
* Consent term signed;

Exclusion Criteria:

* Less than three oocytes for fertilization.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
day three good quality embryo rate | 64-67 hours
  day three A/B embryos

SECONDARY OUTCOMES:
fertilization | 16-18 hours
  presence of 2 pronuclei and 2 polar bodies

CONTACTS AND LOCATIONS:
Overall Officials: João Sabino Cunha Filho, PhD, Study Director — Hospital de Clínicas de Porto Alegre
Locations (1):
- Insemine, Porto Alegre, Rio Grande do Sul, Brazil